CLINICAL TRIAL: NCT04494516
Title: A Qualitative Study to Optimize a Community-Based Pediatric TB/HIV Prevention Intervention and Implementation Strategy
Brief Title: Qualitative Understanding of Community TB Services Pre and Post the CHIP-TB Trial
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: UNITAID (Other); Aurum Institute (Other); KNCV Tuberculosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00237243
Record Dates: First submitted 2020-07-27; First posted 2020-07-31 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Tuberculosis Infection; Tuberculosis Prevention
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-trial: This cohort of participants will be recruited preceding evaluation of the community-based pediatric TB prevention intervention (CHIP-TB; NCT04369326) to assist with design of the intervention and implementation strategy. Participants will include four stakeholder groups including: (1) policy makers, program managers, (2) nurse and physician clinicians, (3) community health team members, and (4) caregivers of child contacts from both South African and Ethiopian sites.
- Post-trial: This cohort of participants will be recruited after evaluation of the community-based pediatric TB prevention intervention (CHIP-TB; NCT04369326) to assist with future scale up and dissemination of the intervention. Participants will include four stakeholder groups including: (1) policy makers, program managers, (2) nurse and physician clinicians, (3) community health team members, and (4) caregivers of child contacts from both South African and Ethiopian sites.

SUMMARY:
This qualitative study is designed to elicit the perspectives of relevant stakeholders to adapt a community-based TB/HIV intervention aimed on providing home-based TB prevention treatment (TPT) initiation for child TB contacts, to design its implementation strategy and, post intervention, to assess lessons learned for future scale up. Participants will include policy makers and health system managers, nurse and physician providers, community health team members, and child caregivers of TB-exposed children. Stakeholders will be asked to participate in two interviews, one prior to the cluster randomized trial assessing this intervention and one after the cluster randomized trial. Trained interviewers will conduct 1-hour semi-structured in-depth interviews that will be audio-recorded, translated and transcribed for thematic analysis using a priori and emergent domains of interest. Free-listing, ranking exercises and cultural consensus will be used to identify context-specific intervention adaptations and implementation strategies.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a top 10 cause of child mortality in sub-Saharan Africa. Short-course combination TB preventive therapy (TPT) regimens are highly effective with high completion rates and therefore hold promise to reduce the 1 million pediatric TB patients and 233,000 child TB deaths annually. TPT effectiveness requires improvement in access to pediatric TB preventive care. The World Health Organization (WHO) estimates only 23% of the 1.3 million TB-exposed children under 5 years old initiated TPT in 2017. The investigators' previous data suggest 50-75% of TB-exposed children under 5 years old fail to be either identified or linked to TB preventive care. Children under 5 years are at exceptionally high risk of TB disease due to not only immature immune systems, but also HIV infection and HIV exposure. Guidelines have long recommended TPT for children under 5 years, but have recently been expanded to children under 15 years. Developing and testing innovative health care delivery models to accompany new WHO-endorsed short-course combination TPT regimens is essential to reduce TB-associated global child morbidity and mortality.

Integrated community case management (iCCM) is a cost-effective intervention that increases child survival by bringing curative therapies to at risk children in the community. Recently, algorithms for screening pediatric patients with household exposure to TB have been simplified to include symptom screening only, eliminating costly laboratory and radiographic evaluations that are barriers to treatment and do not improve sensitivity and specificity of the assessment. The CHIP-TB Trial plans to assess whether integrated community-based pediatric TB/HIV prevention services is feasible, acceptable and effective in increasing TPT uptake among child TB contacts under 15 years in a cluster-randomized trial in South Africa and Ethiopia, two high-burden, resource-limited settings.

Nested within this larger trial, the investigators will use qualitative research to (1) describe the social context in which the community health teams perform the team's duties, (2) make context-specific adaptations to the intervention to maximize its effectiveness, (3) define a context-specific implementation strategy and evaluation plan, and (4) learn important lessons for the future scale up and dissemination of the community-based intervention.

The investigators will conduct 10-15 paired semi-structured individual in-depth interviews (IDI) for each of the four key stakeholder groups: (1) caregivers of TB-exposed children, (2) community health team members, (3) clinic-based nurse and clinic or hospital-based physician providers, and (4) health system managers and policy makers, for a total of ~120 IDIs (~60 in South Africa and ~60 in Ethiopia) both pre and post trial. Before the intervention the investigators will conduct a one-hour interview that will explore the inner setting of the community health team's environment from each stakeholder perspective and will develop and decide upon key intervention adaptations and implementation strategies for the community-based TB/HIV prevention program that will be assessed with a one-year cluster-randomized trial. Upon trial completion, the investigators will conduct another 10-15 semi-structured IDIs with each stakeholder group in each country (total ~120 IDIs) to identify key facilitators and barriers to the implementation. Thematic content analysis with an inductive approach will be used to analyze transcripts for both a priori and emergent domains of interest. A coding scheme will be adapted from Consolidated Framework for Implementation Research (CFIR) constructs. Free listing, ranking, and cultural consensus will be used to identify intervention adaptations and implementation strategies that are context specific. The investigators will use Smith's Saliency Index to analyze the free listed data, mean rank order to assess ranking exercises, and the Eigenvalue to evaluate consensus across groups all using the ANTHROPAC ® 4.0 software.

ELIGIBILITY:
Inclusion Criteria for Interview 1:

* Adult caregiver (18 years of age or older) of a child (<15 years of age) who was exposed to TB in the last two years where at least one child was evaluated for and offered either TB preventive therapy or TB treatment.

or

* Community health team members from one of the Ethiopian or South African clinics in which the CHIP-TB trial will be conducted.

or

* TB nurse from one of the 16 Ethiopian or South African clinics in which the study will be conducted

or

* Pediatrician or medical officer working in pediatrics at the relevant Ethiopian or South African District Hospital who sees outpatient pediatric consultations including TB-exposed children

or

* Program manager or policy maker in the relevant Ethiopian or South African district or provincial office who manages TB, PMTCT, and/or other pediatric programming

Exclusion Criteria for Interview 1:

* Any adult caregivers, community health team members, TB nurses, medical officers or pediatricians, program managers or policy makers who are unable or unwilling to provide informed consent for both the interview and audio-recording

Inclusion Criteria for Interview 2:

* Any community health team members, TB nurses, medical officers or pediatricians, program managers or policy makers who participated in the program for at least 3 months
* Any adult caregiver whose child participated in the community-based TB prevention program

Exclusion Criteria for Interview 2:

* Any adult caregivers, community health team members, TB nurses, medical officers or pediatricians, program managers or policy makers who are unable or unwilling to provide informed consent for both the interview and audio-recording

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include key stakeholders from the target communities in South Africa (Ekurhuleni, Gauteng Province) and Ethiopia (East Shewa Zone of the Oromia regional state), including caregivers of TB-exposed children, community health teams including nurses and community health workers, clinic-based nurse and clinic/hospital-based physician providers, program managers and policy makers.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Perception of intervention adaptations as assessed by an in-depth interview | Within six months prior to CHIP-TB trial initiation
  In-depth, semi-structured interviews will explore perceptions of context-specific adaptations to the community-based TB prevention intervention needed for success.
Perception of implementation strategies as assessed by an in-depth interview | Within six months prior to CHIP-TB trial initiation
  In-depth, semi-structured interviews will explore perceptions of context-specific implementation strategies for the community-based TB prevention intervention needed for success.
Perception of the social context of the community-based health teams as assessed by an in-depth interview | Within six months prior to CHIP-TB trial initiation
  In-depth, semi-structured interviews will explore the social context and inner setting of the community health teams.
Perception of the lessons learned as assessed by an in-depth interview | Within four months after CHIP-TB Trial completion
  In-depth, semi-structured interviews will explore lessons learned for the future scale up and dissemination of the community-based TB prevention intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Salazar-Austin, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- KNCV Tuberculosis Foundation, Addis Ababa, Ethiopia
- The Aurum Institute, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salazar-Austin N, Bergman AJ, Mulder C, Tudor C, Mulatu F, Conradie G, Chaisson RE, Golub JE, Churchyard G, Bedru A, Kerrigan D. Improving access to tuberculosis preventive treatment for children in Ethiopia: designing a home-based contact management intervention for the CHIP-TB trial through formative research. BMC Health Serv Res. 2024 Sep 10;24(1):1043. doi: 10.1186/s12913-024-11451-9. PMID 39252005